CLINICAL TRIAL: NCT05220540
Title: Retrospective Analysis of Balloon Expandable Covered Stenting in the Common Femoral Artery
Acronym: BEST-CFA
Status: Completed | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Csaba Csobay-Novák MD PhD, Head of Noninvasive Imaging, Semmelweis University Heart and Vascular Center
Other Study IDs: AFC2022
Record Dates: First submitted 2022-01-18; First posted 2022-02-02 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: Vascular Complications
Keywords: covered stent; bleeding; closure device; pseudoaneurysm; stenosis; stent fracture
MeSH Terms: conditions — Hemorrhage; Aneurysm, False; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of balloon expandable covered stenting of access complications, stenoses or pseudoaneurysms of the common femoral access.

DETAILED DESCRIPTION:
In the past decades, there has been a paradigm shift in the field of vascular surgery, with endovascular interventions replacing traditional open surgical procedures on an increasing scale. Most of these interventions are performed via the femoral artery. Even with modern percutaneous vascular closure devices, interventional laboratories report a high incidence of vascular complications, most commonly bleeding. Interventional procedures are gaining ground as an alternative to surgery. Having regard to the fact that femoral arteries are in constant motion due to their location and are subject to intense bending forces, the long-term durability of stents has been questioned in the absence of long-term follow-up data. There is currently no broad consensus on the strategy of care for vascular complications, and overall the decision is left to the discretion of the interventionalist, largely determined by the available local resources and infrastructure. The use of covered stents is an option for endovascular treatment of the complications: the self expanding nitinol framed stent graft with polytetrafluoroethylene (PTFE) coating and the cobalt-chrome framed, also PTFE coated balloon expandable stent. The main aim of this research is to analyse the short- and long-term outcome of these alternatives.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* intervention from the left or right common femoral artery
* access complication treated by balloon expandable covered stent(s) or common femoral artery disease treated by balloon-expandable covered stent(s)

Exclusion criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing either transcathether aortic valve repair (TAVR), endovascular aortic repair (EVAR) or thoracic endovascular aortic repair (TEVAR) via percutaneous femoral access resulting in access site complication, or patients who undergo endovascular therapy of common femoral artery disease, managed by balloon-expandable covered stent(s).
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Primary patency rate | 1 year
  Number of patent common femoral arteries at one year
Reintervention rate | 1 year
  Number of reinterventions on the treated vessels
Amputation rate | 1 year
  Number of amputations at the side of the treated common femoral artery

SECONDARY OUTCOMES:
Restenosis rate | 1 year
  Number of significant (peak systolic velocity ratio > 2,4) restenoses found at one year
Walking disturbance rate | 1 year
  Number of any new onset walking impairment

CONTACTS AND LOCATIONS:
Overall Officials: Csaba Csobay-Novák, MD, PhD, Principal Investigator — Semmelweis University Heart and Vascular Center
Locations (3):
- Hungary (3):
  - University of Szeged, Albert Szent-Györgyi Health Center, Second Department of Medicine and Cardiology Centre, Szeged, Csongrád-Csanád
  - Gottsegen National Cardiovascular Center, Budapest
  - Semmelweis University Heart and Vascular Center, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox T, Blair L, Huntington C, Lincourt A, Sing R, Heniford BT. Systematic Review of Randomized Controlled Trials Comparing Manual Compression to Vascular Closure Devices for Diagnostic and Therapeutic Arterial Procedures. Surg Technol Int. 2015 Nov;27:32-44. PMID 26680377
- [Background] Heger T, Strauss S, Blessing E, Andrassy M, Erbel C, Muller OJ, Chorianopoulos E, Pleger S, Leuschner F, Korosoglou G, Bekeredjian R, Katus HA, Vogel B. Short and long-term results after endovascular management of vascular complications during transfemoral aortic valve implantation. Acta Cardiol. 2017 Aug;72(4):474-482. doi: 10.1080/00015385.2017.1335455. Epub 2017 Jul 14. PMID 28705072
- [Background] Barbash IM, Barbanti M, Webb J, Molina-Martin De Nicolas J, Abramowitz Y, Latib A, Nguyen C, Deuschl F, Segev A, Sideris K, Buccheri S, Simonato M, Rosa FD, Tamburino C, Jilaihawi H, Miyazaki T, Himbert D, Schofer N, Guetta V, Bleiziffer S, Tchetche D, Imme S, Makkar RR, Vahanian A, Treede H, Lange R, Colombo A, Dvir D. Comparison of vascular closure devices for access site closure after transfemoral aortic valve implantation. Eur Heart J. 2015 Dec 14;36(47):3370-9. doi: 10.1093/eurheartj/ehv417. Epub 2015 Aug 26. PMID 26314688
- [Background] Schwartz BG, Burstein S, Economides C, Kloner RA, Shavelle DM, Mayeda GS. Review of vascular closure devices. J Invasive Cardiol. 2010 Dec;22(12):599-607. PMID 21127366
- [Background] Sekhar A, Sutton BS, Raheja P, Mohsen A, Anggelis E, Anggelis CN, Keith MC, Dawn B, Straton S, Flaherty MP. Femoral arterial closure using ProGlide(R) is more efficacious and cost-effective when ambulating early following cardiac catheterization. Int J Cardiol Heart Vasc. 2016 Oct 11;13:6-13. doi: 10.1016/j.ijcha.2016.09.002. eCollection 2016 Dec. PMID 28616553
- [Background] Nelson PR, Kracjer Z, Kansal N, Rao V, Bianchi C, Hashemi H, Jones P, Bacharach JM. A multicenter, randomized, controlled trial of totally percutaneous access versus open femoral exposure for endovascular aortic aneurysm repair (the PEVAR trial). J Vasc Surg. 2014 May;59(5):1181-93. doi: 10.1016/j.jvs.2013.10.101. Epub 2014 Jan 17. PMID 24440678
- [Background] Seeger J, Gonska B, Rodewald C, Rottbauer W, Wohrle J. Impact of suture mediated femoral access site closure with the Prostar XL compared to the ProGlide system on outcome in transfemoral aortic valve implantation. Int J Cardiol. 2016 Nov 15;223:564-567. doi: 10.1016/j.ijcard.2016.08.193. Epub 2016 Aug 17. PMID 27561160
- [Background] Durmus G, Belen E, Bayyigit A, Can MM. Comparison of Complication and Success Rates of ProGlide Closure Device in Patients Undergoing TAVI and Endovascular Aneurysm Repair. Biomed Res Int. 2018 Aug 9;2018:2687862. doi: 10.1155/2018/2687862. eCollection 2018. PMID 30175119
- [Background] Franco CD, Goldsmith J, Veith FJ, Calligaro KD, Gupta SK, Wengerter KR. Management of arterial injuries produced by percutaneous femoral procedures. Surgery. 1993 Apr;113(4):419-25. PMID 8456398
- [Background] Tsetis D. Endovascular treatment of complications of femoral arterial access. Cardiovasc Intervent Radiol. 2010 Jun;33(3):457-68. doi: 10.1007/s00270-010-9820-3. Epub 2010 Feb 17. PMID 20162284
- [Derived] Szentivanyi A, Borzsak S, Suvegh A, Berczi A, Szucsborus T, Ruzsa Z, Fontos G, Szalay CI, Papp R, Molnar L, Csobay-Novak C. Midterm Outcome of Balloon-Expandable Covered Stenting of Femoral Access Site Complications. J Clin Med. 2024 Oct 31;13(21):6550. doi: 10.3390/jcm13216550. PMID 39518689